CLINICAL TRIAL: NCT04783870
Title: Effect of Dapagliflozin on Left Ventricular Remodeling in Patients With Acute Myocardial Infarction
Brief Title: Effect of Dapagliflozin on LV Remodeling Post AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Eduardo Almeida Gutiérrez, MD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F-2020-3604-035
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will receive either Dapagliflozin or Placebo. They will not know which arm they have been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg PO QD
  Interventions: Drug: Dapagliflozin
- Control (Placebo Comparator): Placebo PO QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg PO QD
  Arms: Dapagliflozin
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
The overall hypothesis of the study is that Dapagliflozin will reduce left ventricular remodeling in patients who have had a myocardial infarction.

DETAILED DESCRIPTION:
In patients with heart failure, with or without diabetes, SGLT2i have shown to decrease remodeling. However, this has not been tested in patients following an acute myocardial infarction.

Acute myocardial infarction is serious condition with increasing incidence across the world. Following treatment, a reasonable amount of patients develop remodeling of the left ventricle, which is associated with worse prognosis. This occurs despite patients are treated with GDMT.

Dapagliflozin is an SGLT2i with biological plausibility to decrease left ventricular remodeling following acute myocardial infarction. In the present study, researchers will test the hypothesis that Dapagliflozin will reduce left ventricular remodeling in patients who have had a myocardial infarction (less than 7 days). This will be a randomized, single-blind, placebo controlled trial. The primary endpoint will be the change in end-diastolic and end-systolic left ventricular volumes from baseline to the end of the intervention (6 months). We will include patients with acute myocardial infarction who have been treated with primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction treated within the 24 hours of beginning of symptoms
* Signed informed consent
* SBP > 90 mmHg
* Age >= 18 years

Exclusion Criteria:

* Glomerular Filtration Rate < 30 ml/min/1.73 m2.
* Pregnant or lactating woman
* Cancer or life-threatening condition
* Use of continuous parental inotropic agents
* Psychiatric disease incompatible with being in study.
* Any contraindication to MRI procedures.
* Any other medical or physical condition considered to be inappropriate by a study physician
* Scheduled for a PCI or CABG within the next 6 months
* Hemodynamic unstability
* Currently on any SGLT2i
* One or more episodes of severe hypoglicemia
* Acute urinary or genital infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular remodeling | 6 months
  Changes in end-diastolic and end-systolic left ventricular volumes

SECONDARY OUTCOMES:
Natriuretic peptides | 6 months
  Change in natriuretic peptide
Quality of life assessed with KCCQ | 6 months
  Change in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Ivey-Miranda, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Cardiología, Centro Médico Nacional Siglo XXI, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared only to researches with extensive research. These will be analyzed on case-by-case basis.
Supporting Information: Study Protocol, CSR
Time Frame: After the study termination
Access Criteria: IPD will be shared only to researches with extensive research. These will be analyzed on case-by-case basis.